CLINICAL TRIAL: NCT00669344
Title: A 24-week Prospective, Double Blind, Randomized, Placebo-controlled Pilot Study of 9 mg/Day Rivastigmine in Patients With Vascular Cognitive Impairment Not Dementia to Evaluate Efficacy, Safety and Tolerability in Asian Patients
Brief Title: RIVastigmine In Vascular cognitivE Impairment
Acronym: RIVIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Novartis (Industry); National Neuroscience Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CENA713BSG01
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Cognitive Impairment
Keywords: cognition; stroke; VCI; VCIND; Cognitive Impairment, No Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Stroke | interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- II (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- I (Experimental): Rivastigmine
  Interventions: Drug: Exelon (rivastigmine)

INTERVENTIONS:
Drug: Exelon (rivastigmine) — Capsules, twice daily orally. Dosage starts at 1.5mg bis diem to 4.5mg bis diem.
  Arms: I
Drug: Placebo — Capsule, twice daily orally. Dosage starts at 1.5mg bis diem to 4.5mg bis diem.
  Arms: II

SUMMARY:
The study is a 24-week prospective, double blind, randomized, placebo-controlled pilot study of 9 mg / day Rivastigmine in patients with Vascular Cognitive Impairment Not Dementia (CIND) to evaluate efficacy, safety and tolerability in Asian patients. The hypothesis is that patients receiving Rivastigmine would improve in executive functioning domains.

DETAILED DESCRIPTION:
Methodology: This is a 24-week, double blind, randomized, placebo-controlled pilot study of 9 mg / day Rivastigmine in patients with Cognitive Impairment Not Dementia due to cerebrovascular disease.

During the screening period, patients will be evaluated for CIND by means of neuropsychological tests establishing cognitive impairment following stroke or resulting from subcortical ischemic vascular disease (diagnosed by MRI) AND exclusion of dementia by DSM-IV criteria. At baseline, eligible patients will be evaluated for additional inclusion/exclusion criteria, vital signs, MMSE, Ten Point Clock Test, Colour Trails Test 1 & 2, ADAS-Cog, Cognitive Battery, Frontal Assessment Battery (FAB), Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) scale for mild cognitive impairment (MCI), Neuropsychiatric Inventory (NPI), Geriatric Depression Scale (GDS) and past/coexistent medical conditions. Laboratory examinations and ECGs will be evaluated at screening and week 24.

Patients will be evaluated every 4 weeks for 12 weeks at which time dose increases will be made and vital signs will be evaluated. At Week 12, cognitive and functional measures will be evaluated including the Ten Point Clock Test, Colour Trails Test 1 & 2, ADAS-Cog, Cognitive Battery, FAB, ADL Scale for MCI, and NPI and GDS will be evaluated. At week 16 and week 20, telephone calls will be made to patients and caregivers to ascertain compliance. At Week 24, cognitive and functional measures will be evaluated including the Ten Point Clock Test, Colour Trails Test 1 & 2, ADAS-Cog, Cognitive Battery, FAB, ADL Scale for MCI, and NPI and GDS will be evaluated.

Patients will be receiving a bottle of trial drug at appropriate titration dose every 4 weeks during titration phase starting from rivastigmine/placebo 1.5mg bd daily. During maintenance phase / at week 12, patients will be given 3 bottles of trial drug at the appropriate maintenance dose.

Adverse events and serious adverse events will be captured at every visit. In addition, patients who discontinue the study will be followed for safety evaluations through 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients, age 55-85
* outpatients, living with a caregiver
* Rankin score <=3
* Diagnosis of Cognitive Impairment Not Dementia due to cerebrovascular disease
* Post-stroke cognitive impairment
* Cognitive impairment documented by neuropsychological evaluation within 6 months of index stroke

Exclusion Criteria:

* Advanced, severe, and unstable disease of any type that may interfere with the efficacy evaluations or put the subject at special risk
* A current diagnosis of active uncontrolled seizure disorder
* A current diagnosis of active peptic ulceration
* A current diagnosis of severe and unstable cardiovascular disease
* A current diagnosis of sick-sinus syndrome or conduction deficits (sino-atrial block, atrioventricular block)
* A current diagnosis of unstable angina
* MI within the last 6 months
* DSM IV current diagnosis of dementia
* DSM IV current diagnosis of major depression (patients may be included if currently being treated on an antidepressant and stabilized after 3 months)
* A disability that may prevent the subject from completing all study requirements (e.g. blindness, deafness, severe language difficulty)
* A known exaggerated pharmacological sensitivity or hypersensitivity to acetylcholinesterase inhibitors or to other cholinergic compounds
* Ingestion of any of the following:
* an investigational drug in the past four weeks
* metrifonate in the last 3 months
* a drug or treatment known to cause major organ system toxicity during the past four weeks
* other cholinergic drugs (eg succinylcholine type muscle relaxants) during the past two weeks
* anticholinergics prior to baseline
* acetylcholinesterase inhibitors in the past 3 months
* Women of childbearing potential

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the comparative change from baseline between treatment and placebo arms in the Ten Point Clock Drawing Test as well as Color Trails 1 and 2. | week 24

SECONDARY OUTCOMES:
To evaluate the comparative change from baseline between treatment and placebo on cognitive function | week 24
To evaluate the comparative change from baseline between treatment and placebo on activities of daily living | week 24
To evaluate the comparative change from baseline between treatment and placebo on behavior and depression | week 24
To evaluate the safety and tolerability of treatment in comparison to placebo | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Eng King Tan, FAMS, Principal Investigator — National Neuroscience Institute, Singapore General Hospital Campus
Locations (1):
- Singapore General Hospital, Singapore, Singapore